CLINICAL TRIAL: NCT06253000
Title: Comparative Analysis of Radiofrequency and Cryoablation of the Posterior Wall of the Left Atrium in Patients With Persistent Atrial Fibrillation
Brief Title: Radiofrequency and Cryoablation of the Posterior Wall of the Left Atrium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bakulev Scientific Center of Cardiovascular Surgery (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #4.10.11.2022
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Acute Cerebrovascular Accident; Transient Ischemic Attack; Death; Atrial Fibrillation Recurrent
Keywords: atrial fibrillation; radiofrequency ablation; cryoablation; left atrium; the posterior wall of the left atrium; atrial remodeling
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Death; Atrial Fibrillation; Atrial Remodeling | interventions — Cryosurgery; Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: A randomized double-blind controlled trial in two groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoablation (Active Comparator): Cryoablation of the mouths of the pulmonary veins and the posterior wall of the left atrium.
  Interventions: Procedure: Cryoablation
- Radiofrequency ablation (Active Comparator): Radiofrequency ablation of pulmonary veins according to the "box isolation" type using a non-fluoroscopic navigation system.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Cryoablation — Cryoablation of the mouths of the pulmonary veins and the posterior wall of the left atrium.
  Arms: Cryoablation
Procedure: Radiofrequency ablation — Radiofrequency ablation of pulmonary veins according to the "box isolation" type using a non-fluoroscopic navigation system.
  Arms: Radiofrequency ablation

SUMMARY:
Atrial fibrillation (AF) is the cause of 20% of strokes, and the risk of stroke in a person suffering from this arrhythmia increases by 5 times. Ischemic stroke in patients with AF is often fatal and, compared with stroke of other etiology, leads to the most pronounced disability and more often recurs. Accordingly, the risk of death in patients with AF-related stroke is 2 times higher, and treatment costs increase 1.5 times.

The main interventional method of treating AF, available in most medical institutions, is the use of radio frequency and/or cryoenergy to eliminate destructive damage to the left atrium (LA).

The aim of this study is to compare two different interventional methods and identify predictors of recurrence in patients with persistent and long-term AF.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old;
* Atrial fibrillation resistant to antiarrhythmic therapy;
* Persistent and long-persisting form of atrial fibrillation;
* The patient's consent to participate in the study.

Exclusion Criteria:

* Age under 18 and over 80 years old;
* The presence of another cardiac pathology requiring surgical treatment;
* Congenital heart defects;
* Previous "open" cardiac surgery;
* Bone marrow diseases;
* Pathology of the blood coagulation system;
* The left ventricular ejection fraction is less than 40%;
* Moderate to severe renal insufficiency (creatinine clearance <50 ml/min);
* Drug-resistant hypertension (despite hypotensive therapy);
* Organically altered mitral valve;
* There are reasons to assume that the patient will not show up for subsequent visits (control points of the study) for various reasons;
* The patient's participation in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cerebral events | From the date of ablation until the date of the event, assessed up to 24 months.
  The number of patients who had a stroke or acute cerebrovascular accident or a transient ischemic attack within 24 months after ablation.

SECONDARY OUTCOMES:
Hospital mortality | From the date of ablation until the date of death, assessed up to 5 days.
  The number of patients who died in the hospital.
Non-lethal events | From the date of ablation to the date of any of the listed events, assessed up to 5 days.
  Number of participants with non-lethal events. The main hospital non-lethal events (bleeding, tamponade, perforation of the walls of the heart, damage to the esophagus).
Recurrence of AF | From the date of ablation until the date of recurrent atrial fibrillation, assessed up to 24 months.
  The number of patients with recurrent atrial fibrillation after surgery.
Long-term mortality | From the date of ablation until the date of death, assessed up to 24 months.
  The number of patients who died during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Filatov, Principal Investigator — Bakulev Scientific Center for Cardiovascular Surgery
Locations (1):
- Bakulev National Medical Research Center for Cardiovascular Surgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No